CLINICAL TRIAL: NCT05373667
Title: A Prospective Clinical Study to Assess the Spinal Cord Stimulation System in the Treatment of Chronic Pelvic Pain
Acronym: SCS/CPP
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Europainclinics z.ú. (Other)
Collaborators: National Hospital for Neurology and Neurosurgery, London (Unknown)
Responsible Party: Sponsor
Other Study IDs: NSM 1-129/2021
Record Dates: First submitted 2022-05-04; First posted 2022-05-13 (Actual); Last update posted 2022-05-13 (Actual); Status verified 2022-05

CONDITIONS: Pelvic Pain
Keywords: Spinal cord Stimulation, Pelvic Pain
MeSH Terms: conditions — Pelvic Pain | interventions — Spinal Cord Stimulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Spinal Cord Stimulation (SCS) — Spinal Cord Stimulation (SCS) - High Frequency at 10 kHz

SUMMARY:
Prospective observational assessment of the efficacy of Spinal Cord Stimulation (SCS) treatment in patients with neuropathic pelvic pain.

DETAILED DESCRIPTION:
The objective of a clinical trial is an assessment of the efficacy of Spinal Cord Stimulation (SCS) treatment in patients with localized (not widespread pain), predominant neuropathic pelvic pain neuropathic pain (determined by PAIN-DETECT and rule out musculature pain).

Etiologies of CPP to be studied include but not limited to vulvodynia, perineal pain, perianal pain, bladder pain syndrome, and pelvic pain resulting from colorectal procedures. Medical review of the subjects will be done by a multidisciplinary team consisting of urologists/ gynecologists, interventional pain physicians, and psychiatrists.

Enrolled centers are National Hospital For Neurology and Neurosurgery in London in the United Kingdom, EuroPainClinics® with centers in Bratislava, Košice, and Bardejov in the Slovac republic and also EuroPainClinics® with centers Praha, Brno, Ostrava, and Hradec Kralove in the Czech republic.

Lead placement:

To be determined as a function of pain distribution. Lead placement will be either retrograde or anterograde determined by the investigator.

Study Duration:

The expected duration of this study is approximately 12 months. Enrollment is expected to last 6 months, with subjects followed up to a 12 month period following permanent implant. The time commitment for a subject to complete the study is approximately 13 months; consisting of Baseline assessments, and last follow-up at 12 months.

Study Design:

This is a single-center, single-arm, prospective, observational post-market study to assess the safety and effectiveness of the Senza System in subjects with chronic pelvic pain. Subjects are acting as his/her own control. Data at follow-up visits will be compared to the subjects' baseline data.

Study Objective:

The objective of this observational study is to assess the safety and effectiveness of the Spinal cord stimulation, in the treatment of Chronic Pelvic Pain at the study follow-up visits at 1, 3, 6, 9 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* 1. Have a clinical diagnosis of chronic predominant pelvic pain as determined by a multidisciplinary study team.

  2. Score 13 or greater in PainDETECT questionnaire 3. 4. Have been refractory to conservative therapy for a minimum of 3 months, including assessment of at least 2 different classes of medications.

  5. Average pain intensity (over the last 7 days) of ≥ 5 out 10 cm on the Visual Analog Scale (VAS) in the primary area of pain at enrollment (in accordance with the NICE guidelines).

  6. Have stable neurological status measured by motor, sensory and reflex function as determined by the investigator.

  7. Be on stable pain medications, as determined by the Investigator, for at least 28 days prior to assessing pain intensity as described in inclusion criterion.

  8. Be 18 years of age or older at the time of enrollment. 9. Be an appropriate candidate for the surgical procedures required in this study based on the clinical judgment of the implanting physician.

  10. Be capable of subjective evaluation, able to read and understand written questionnaires, and are able to read, understand and sign the written inform consent.

  11. Be willing and capable of giving informed consent. 12. Be willing and able to comply with study-related requirements, procedures, and visits.

  13. Have adequate cognitive ability to use a patient programmer and recharger as determined by the Investigator

Exclusion Criteria:

1. Have a medical condition or pain in other area(s), not intended to be treated with SCS, that could interfere with study procedures, accurate pain reporting, and/or confound evaluation of study endpoints, as determined by the investigator (such as primary headache diagnosis or fibromyalgia).
2. Have a current diagnosis of a progressive neurological disease such a multiple sclerosis, chronic inflammatory demyelinating polyneuropathy, rapidly progressive arachnoiditis, brain or spinal cord tumor, central deafferentation syndrome, Complex regional Pain Syndrome, acute herniating disc, severe spinal stenosis and brachial plexus injury as determined by the investigator.
3. Have a current diagnosis or condition such as a coagulation disorder, bleeding diathesis, platelet dysfunction, progressive peripheral vascular disease or uncontrolled diabetes mellitus that presents excess risk for performing the procedure as determined clinically by the investigator.
4. Significant stenosis, objective evidence of epidural scarring and/or any signs or symptoms of myelopathy as determined by MRI conducted within the past 12 months.
5. Have a clinical diagnosis of unstable mental health condition or severe depression [request input on this exclusion criteria from the psychologist] including suicidal ideation.
6. Be benefitting within from an interventional procedure and/or surgery to treat chronic pelvic pain (Subjects should be enrolled at least 30 days from last benefit).
7. Have an existing drug pump and/or another active implantable device such as a pacemaker.
8. Have failed other neuromodulation therapies including traditional SCS, peripheral nerve stimulation or dorsal root ganglion stimulation.
9. Have metastatic malignant disease or active local malignant disease.
10. Have a life expectancy of less than 1 year.
11. Have an active systemic or local infection at the anticipated needle entry site.
12. Be pregnant or plan to become pregnant during the study (participants of child-bearing potential that are sexually active must use a reliable form of birth control).
13. Are currently nursing (if female).
14. Have been immunocompromised.
15. Have been known to be allergic or have shown hypersensitivity to any materials of the neurostimulation system which come in contact with the body.
16. Have within 6 months of enrollment a significant untreated addiction to dependency producing medications or have been a substance abuser (including opioids, benzodiazepines, alcohol and illicit drugs).
17. Be concomitantly participating in another clinical study.
18. Be involved in an injury claim under current litigation.
19. Have a pending or approved worker's compensation claim.
20. Presence of pelvic tumor including benign.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with chronic pelvic pain
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2023-08-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Visual analog scale | 1 month follow-up
Visual analog scale | 3 month follow-up
Visual analog scale | 6 month follow-up
Visual analog scale | 9 month follow-up
Visual analog scale | 12 month follow-up
Pain Disability Index | 1 month follow-up
Pain Disability Index | 3 month follow-up
Pain Disability Index | 6 month follow-up
Pain Disability Index | 9 month follow-up
Pain Disability Index | 12 month follow-up
McGill Pain questionnaire (SF-MPQ-2) | 1 month follow-up
McGill Pain questionnaire (SF-MPQ-2) | 3 month follow-up
McGill Pain questionnaire (SF-MPQ-2) | 6 month follow-up
McGill Pain questionnaire (SF-MPQ-2) | 9 month follow-up
McGill Pain questionnaire (SF-MPQ-2) | 12 month follow-up
European Quality of Life-5 Dimensions (EQ-5D-5L) | 1 month follow-up
European Quality of Life-5 Dimensions (EQ-5D-5L) | 3 month follow-up
European Quality of Life-5 Dimensions (EQ-5D-5L) | 6 month follow-up
European Quality of Life-5 Dimensions (EQ-5D-5L) | 9 month follow-up
European Quality of Life-5 Dimensions (EQ-5D-5L) | 12 month follow-up
Short Form 12-Item Survey on Health (SF-12) | 1 month follow-up
Short Form 12-Item Survey on Health (SF-12) | 3 month follow-up
Short Form 12-Item Survey on Health (SF-12) | 6 month follow-up
Short Form 12-Item Survey on Health (SF-12) | 9 month follow-up
Short Form 12-Item Survey on Health (SF-12) | 12 month follow-up

SECONDARY OUTCOMES:
Neurologic status | 6 month follow-up
  includes motor, sensory and reflex functions, which will be characterized as improved, maintained, or a deficit as compared with baseline status as follows:
  1. A clinically meaningful neurological and physical status improvement is defined as a significant persistent improvement in neurological function that impacts subject's well-being is attributable to a neurological finding; and is new or improved as compared with the baseline assessment.
  2. A clinically meaningful neurological deficit is defined as a stimulation-related significant persistent abnormality in neurological function that impacts subject's well-being is attributable to a neurological finding; and is new or worsened as compared with the baseline assessment.
  3. If neither a clinically meaningful neurological improvement nor a clinically meaningful neurological deficit is observed, then neurologic status is maintained.
Neurologic status | 12 month follow-up
  includes motor, sensory and reflex functions, which will be characterized as improved, maintained, or a deficit as compared with baseline status as follows:
  1. A clinically meaningful neurological and physical status improvement is defined as a significant persistent improvement in neurological function that impacts subject's well-being is attributable to a neurological finding; and is new or improved as compared with the baseline assessment.
  2. A clinically meaningful neurological deficit is defined as a stimulation-related significant persistent abnormality in neurological function that impacts subject's well-being is attributable to a neurological finding; and is new or worsened as compared with the baseline assessment.
  3. If neither a clinically meaningful neurological improvement nor a clinically meaningful neurological deficit is observed, then neurologic status is maintained.
Hospitalizations | 12 month follow-up
  compared to baseline history of previous 12 months
Adverse events | 12 month follow-up
Medication usage | 12 month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Róbert Rapcan, MD, PhD, MBA, FIPP, Study Director — Europainclinics z.ú.; Ladislav Kočan, MD, PhD, Study Chair — Europainclinics z.ú.